CLINICAL TRIAL: NCT01203046
Title: SP1 - Early Short-term Antibiotic Therapy in Penetrating Abdominal Trauma, 3 vs 7 Days
Brief Title: Early Short-term Antibiotic Therapy in Penetrating Abdominal Trauma, 3 vs 7 Days
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Silvia M. Pinango L. (Individual)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Silvia M. Pinango L., Pinango L, Silvia M., Pinango, Silvia M. L., M.D.
Organization: Pinango, Silvia M. L., M.D. (Individual)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SP 01
Record Dates: First submitted 2010-09-14; First posted 2010-09-16 (Estimated); Results first posted 2012-07-26 (Estimated); Last update posted 2012-08-10 (Estimated); Status verified 2012-08

CONDITIONS: SURGICAL SITE INFECTION
Keywords: DURATION OF THERAPY; PENETRATING ABDOMINAL TRAUMA
MeSH Terms: conditions — Surgical Wound Infection | interventions — Ertapenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GROUP A: 7 DAYS ANTIBIOTIC THERAPY (Active Comparator): Ertapenem will be administrated within the first 2 hours of Hospital´s admission and the during the next 7 days after surgery.
  Interventions: Drug: Ertapenem
- GROUP B - 3 DAYS ANTIBIOTIC THERAPY (Experimental): Ertapenem will be administrated within the first 2 hours of Hospital´s admission and during the next 3 days after surgery.
  Interventions: Drug: Ertapenem

INTERVENTIONS:
Drug: Ertapenem — Ertapenem 1 gr endovenous 3 or 7 days
  Other Names: Invanz; Early antibiotic therapy

SUMMARY:
Abdominal penetrating trauma represents a frequent cause of consult into emergency rooms in Venezuela. Accidents and violence at Hospital "Miguel Perez Carreño" along april 2009 were represented by gunshots and stabbing wounds which 8th. and 18th cause for medical attention respectively within a total of 76 cases. Likewise gunshot wounds reach the first cause of morbility into general surgery services with 21 cases and the stabbing wounds the 12th cause with 12 cases within the same period.

Early therapy is defined as the antibiotic dose administrated within the first 12 hours after the trauma. Abdominal cavity contamination by micro-organism is not synonymous of stablished infection, the extension of contamination and intensity of reaction should be enough in order to allow the inflammatory focus developing.

Abdominal cavity needs at least 12 - 24 hours of exposure to the infectious material to allow the stablishment of such infection. Origin and amount of contaminant material influence the size of inoculated bacteria and the speed that infection develops.

There is not an absolute criteria to determine when intrabdominal contamination progress to an established infection. Surgeons decides the must adequated therapy according to clinical history, radiology tests and findings during surgery.

Selected patients for early antibiotic therapy in penetrating abdominal trauma includes those with traumatic intestinal wounds with less than 12 hours of evolution and those with gastroduodenal wounds lesser than 24 hours as well.

There are different antibiotics indicated for intrabdominal infections. Ertapenem is a low resistance carbapenem with a broad spectrum into microbial flora presenting in penetrating abdominal trauma. Its media life and blood therapeutic levels allows the use of an unique dose within the first 24 hours of trauma.

This research protocol has been designed according to established patterns for clinical investigation and our goal is to achieve criteria in decision making about antibiotic administration in patients with penetrating abdominal trauma and evaluate the security of an Early short term antibiotic therapy with Ertapenem 3 days vs 7 days, decreasing hospital costs related to indiscriminate use of antibiotics.

DETAILED DESCRIPTION:
General objectives The object of this research is to evaluated the impact of Early short-term antibiotic therapy with Ertapenem, 3 vs 7 days, upon clinical postoperatory evolution in patients with penetrating abdominal trauma at emergency room of "Miguel Perez Carreño" Hospital

Specific objectives

1. To determine the incidence of postoperatory infectious complications in patients with penetrating abdominal trauma under Early short term antibiotic therapy with Ertapenem.
2. To establish the efficacy of Early short term antibiotic therapy 3 days with Ertapenem versus systematic administration of the same antibiotic up to the 7th day after surgery in order to prevent postoperatory infections.
3. To identify the risk factors that predispose the appearance of infectious complications in patients with penetrating abdominal trauma.

Investigation type This will be a prospective, comparative, double blind, randomized, experimental clinical trial in patients with penetrating abdominal trauma, who attend the emergency room of Dr. "Miguel Perez Carreño" Hospital between February and July 2010.

Therapy. Surgery will be perform within a period no longer than twelve hours since time of trauma. Culture samples from abdominal cavity will be taken during the surgery in order to identify the bacterial prevalence and its sensibility to antibiotics.

Ertapenem will be administrated within the first 2 hours of Hospital´s admission and the next two days after surgery. At day four, patients will be assigned to different groups A or B, according to they entrance number into this trial.

Group A treatment will be continued with Ertapenem until 7th day. Group B antibiotic therapy will be stopped.

Patients follow up will be done during the first 10 days after trauma in two phases:

1. First 7 days patients will be controlled by a daily evaluation and the data will be recorded according to variables in the control sheet (Appendix 3).
2. Patients with evolution as follows, will be treated under medical criteria and cultures results:

   1. Temperature 38,5 °C or higher more than 24 hours within the first 7 postoperatory days.
   2. Sustained WBC count higher than 14,000 or increase after 48 hrs. Postoperatory.
   3. Postoperatory complications such as gastric or intestinal fistula, purulent drainage, intrabdominal abscess.
3. On day 10 a new evaluation of patients will be performed and recorded in the control sheet (Appendix 4).

Evaluation variables. Information will be recorded by full register of standard control sheets which includes: admittance date, medical history number, age, sex, clinical conditions, associated comorbidity, surgical findings, time since trauma, surgery time, and starting time of antibiotic administration (Appendix 1).

Penetrating abdominal trauma scale will be applied in order to determine the seriousness of trauma and its potential general echoes (Appendix 2).

During the postoperatory period the control sheet will include: WBC count, albumin, lymphocyte, local conditions of the surgical wound and penetration site wound at the abdominal wall, complications(Appendix 3).

After patient discharge, they will be appointed and evaluated 10 to 12 days after surgery and the following items will be recorded: local conditions of the surgical wound, and penetration site wound, complications. (Appendix 4).

Data from excluded patients will be recorded by exclusion causes and their evolution (Appendix 5). Result of sample cultures taken during surgery and its antibiogram will be reported (Appendix 6).

Operations plan timetable

1. Problem identification request and project design. October 2009 - Feb 2010.
2. Authorization request to the Bioethics Board of "Dr. Miguel Perez Carreño" Hospital. Feb 2010.
3. Authorization request to the Technical Commission of "Dr. Miguel Perez Carreño" Hospital. Feb 2010
4. Development and execution. Feb Nov - 2010.
5. Data analysis. November 2010.
6. Presentation and introduction for publication.

Data processing analysis.

To establish non-inferiority of the use of the therapy with ertapenem between three days versus 7 days of treatment, was considered a significance level of 5%, 95% confidence interval, a power of 80% and in the group control of 60%, a margin of not less 10% is considered of no clinical importance. For a balanced design of type n1 = n2 r = 1. Still needed 26 patients per group. The period of advance recruitment of patients was 6 months.

Ethical aspects. It will be required and informed consent to individuals whom enter to this study, after explaining to them what is all about, the benefits and the possible risks, they wil be asked for their signatures or the signatures of closest relatives at the entrance time. (Appendix 6).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with penetrating abdominal trauma who attended the emergency room within 12 hours after trauma, admitted to an exploratory laparotomy.
2. Patients aged 12 to 65 years.

Exclusion Criteria:

1. Clinical history of immunologic diseases, cancer, use of immunosuppressors, steroids, malnutrition, morbid obesity.
2. Concomitant pathology at admittance: urinary infections, respiratory infections, hepatitis, viral diseases.
3. Associated open bone fractures.
4. Patients with hemodynamic instability during pre or peroperative.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2010-12; Primary Completion 2010-12 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: SILVIA M. PIÑANGO, MD, Principal Investigator — IVSS Dr. MIGUEL PEREZ CARREÑO HOSPITAL; LUIS R. LEVEL, MD FACS, Study Chair — IVSS Dr. MIGUEL PEREZ CARREÑO HOSPITAL

REFERENCES:
- [Background] Dellinger EP. Antibiotic prophylaxis in trauma: penetrating abdominal injuries and open fractures. Rev Infect Dis. 1991 Sep-Oct;13 Suppl 10:S847-57. doi: 10.1093/clinids/13.supplement_10.s847. PMID 1754794
- [Background] Kirton OC, O'Neill PA, Kestner M, Tortella BJ. Perioperative antibiotic use in high-risk penetrating hollow viscus injury: a prospective randomized, double-blind, placebo-control trial of 24 hours versus 5 days. J Trauma. 2000 Nov;49(5):822-32. doi: 10.1097/00005373-200011000-00006. PMID 11086771
- [Background] Bozorgzadeh A, Pizzi WF, Barie PS, Khaneja SC, LaMaute HR, Mandava N, Richards N, Noorollah H. The duration of antibiotic administration in penetrating abdominal trauma. Am J Surg. 1999 Feb;177(2):125-31. doi: 10.1016/s0002-9610(98)00317-1. PMID 10204554
- [Background] Schnuriger B, Inaba K, Eberle BM, Wu T, Talving P, Bukur M, Belzberg H, Demetriades D. Microbiological profile and antimicrobial susceptibility in surgical site infections following hollow viscus injury. J Gastrointest Surg. 2010 Aug;14(8):1304-10. doi: 10.1007/s11605-010-1231-x. Epub 2010 May 25. PMID 20499202
- [Background] de Lalla F. Antimicrobial chemotherapy in the control of surgical infectious complications. J Chemother. 1999 Dec;11(6):440-5. doi: 10.1179/joc.1999.11.6.440. PMID 10678785
- [Background] Borbone S, Cascone C, Santagati M, Mezzatesta ML, Stefani S. Bactericidal activity of ertapenem against major intra-abdominal pathogens. Int J Antimicrob Agents. 2006 Nov;28(5):396-401. doi: 10.1016/j.ijantimicag.2006.07.018. Epub 2006 Oct 11. PMID 17045463
- [Background] Girgin S, Gedik E, Uysal E, Tacyildiz IH. Independent risk factors of morbidity in penetrating colon injuries. Ulus Travma Acil Cerrahi Derg. 2009 May;15(3):232-8. PMID 19562544
- [Background] Salim A, Teixeira PG, Inaba K, Brown C, Browder T, Demetriades D. Analysis of 178 penetrating stomach and small bowel injuries. World J Surg. 2008 Mar;32(3):471-5. doi: 10.1007/s00268-007-9350-6. PMID 18196326
- [Background] Morales CH, Villegas MI, Villavicencio R, Gonzalez G, Perez LF, Pena AM, Vanegas LE. Intra-abdominal infection in patients with abdominal trauma. Arch Surg. 2004 Dec;139(12):1278-85; discussion 1285. doi: 10.1001/archsurg.139.12.1278. PMID 15611450
- [Background] Oreskovich MR, Dellinger EP, Lennard ES, Wertz M, Carrico CJ, Minshew BH. Duration of preventive antibiotic administration for penetrating abdominal trauma. Arch Surg. 1982 Feb;117(2):200-5. doi: 10.1001/archsurg.1982.01380260068012. PMID 7055433
- [Background] Farre Rovira R, Frasquet Pons I, Ibor Pica JF. [Postoperative complications in malnourished patients: economic impact and predictive value of some nutritional indicators]. Nutr Hosp. 1998 Sep-Oct;13(5):233-9. Spanish. PMID 9830844
- [Background] Scheunemann L, Wazlawik E, Bastos JL, Ristow Cardinal T, Mayumi Nakazora L. Agreement and association between the phase angle and parameters of nutritional status assessment in surgical patients. Nutr Hosp. 2011 May-Jun;26(3):480-7. doi: 10.1590/S0212-16112011000300008. PMID 21892564
- [Background] Pull ter Gunne AF, Skolasky RL, Ross H, van Laarhoven CJ, Cohen DB. Influence of perioperative resuscitation status on postoperative spine surgery complications. Spine J. 2010 Feb;10(2):129-35. doi: 10.1016/j.spinee.2009.10.002. Epub 2009 Nov 14. PMID 19914877
- [Background] Cheadle WG. Risk factors for surgical site infection. Surg Infect (Larchmt). 2006;7 Suppl 1:S7-11. doi: 10.1089/sur.2006.7.s1-7. PMID 16834549

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The data was collected between December 2010 and November 2011 including patients with penetrating abdominal trauma admitted at Dr. Miguel Perez Carreño Hospital emergency room.
Pre-assignment Details: We were behind schedule to start the trial waiting for institutional approve.
Groups:
- GROUP A: 7 DAYS ANTIBIOTIC THERAPY: Ertapenem will be administrated within the first 2 hours of Hospital´s admission and the next two days after surgery. At day four, patients will be assigned to different groups A or B, according to they entrance number into this trial.
  Group A will be treated with Ertapenem during the following four days.
- GROUP B: 3 DAYS ANTIBIOTIC THERAPY: Ertapenem will be administrated within the first 2 hours of Hospital´s admission and the next two days after surgery. At day four, patients will be assigned to different groups A or B, according to they entrance number into this trial.
  Group B will be treated with placebo during the following four days.
Period: Overall Study
Arm/Group | GROUP A: 7 DAYS ANTIBIOTIC THERAPY | GROUP B: 3 DAYS ANTIBIOTIC THERAPY
Started | 28 | 28
Completed | 28 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GROUP A: 7 DAYS ANTIBIOTIC THERAPY | GROUP B: 3 DAYS ANTIBIOTIC THERAPY | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 3 | 10
  Between 18 and 65 years | 21 | 25 | 46
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 26.2857 (9.5450) | 28.5000 (9.8639) | 27.3929 (9.6929)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 26 | 25 | 51
Type of trauma [Number; unit: participants] — To describe the mechanism of penetrating abdominal trauma: Gun shot wound (GSW) or Stab wound (SW)
  participants
    GSW | 24 | 22 | 46
    SW | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Surgical Site Infection
Description: The patients were evaluated up to 10 days with close observation of surgical site. We concluded as surgical site infection when inflammatory signs, purulent discharge, intestinal liquid and aponeurosis disruption was observed.
Time Frame: 10 days
Population: All patients with inflammatory signs, purulent discharge, intestinal liquid and aponeurosis disruption observed at surgical site were included.
Measure: Number; unit: participants
Groups:
- GROUP A: 7 DAYS THERAPY: Ertapenem will be administrated within the first 2 hours of Hospital´s admission and the next two days after surgery. At day four, patients will be assigned to different groups A or B, according to they entrance number into this trial.
  Group A will be treated with Ertapenem during the following four days.
- GROUP B - 3 DAYS THERAPY: Ertapenem will be administrated within the first 2 hours of Hospital´s admission and the next two days after surgery. At day four, patients will be assigned to different groups A or B, according to they entrance number into this trial.
  Group B will be treated with placebo during the following four days.
Arm/Group | GROUP A: 7 DAYS THERAPY | GROUP B - 3 DAYS THERAPY
Number analyzed (Participants) | 28 | 28
participants | 6 | 3
Statistical Analysis 1: Comparison: GROUP A: 7 DAYS THERAPY vs GROUP B - 3 DAYS THERAPY; Test type: Non-Inferiority or Equivalence — It was used for the calculation of statistical power an author of 5% level, it was felt that the difference between the minimum value of non inferiority does not exceed 10%; p < 0.05, Regression, Logistic; Odds Ratio (OR) = 2.65, 95% CI 2-sided [0.35 to 19.83]

2. Primary Outcome: Other Complications
Description: Patients with complications different to surgical site infection.
Time Frame: 10 days
Population: Patients who presented any complication different of surgical site infection after surgery
Measure: Number; unit: participants
Groups:
- GROUP A - 7 DAYS THERAPY: Patients with 7 days therapy
- GROUP B - 3 DAYS THERAPY: Patients with 3 days therapy
Arm/Group | GROUP A - 7 DAYS THERAPY | GROUP B - 3 DAYS THERAPY
Number analyzed (Participants) | 28 | 28
participants | 8 | 5
Statistical Analysis 1: Comparison: GROUP A - 7 DAYS THERAPY vs GROUP B - 3 DAYS THERAPY; Test type: Non-Inferiority or Equivalence — Consider a 5% confidence level, the power of assigned contrast was 80% to detect a difference minima of at least 10% of equivalence between the analyzed groups; p < 0.05, Regression, Logistic; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.21 to 6.51]

ADVERSE EVENTS:
Arm/Group | GROUP A: 7 DAYS ANTIBIOTIC THERAPY | GROUP B: 3 DAYS ANTIBIOTIC THERAPY
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28

LIMITATIONS AND CAVEATS:
Presented limitations because patients with penetrating abdominal trauma usually had associated bone fractures or haemodynamic instability.Identifying other predisposing factors is not reached since the sample size was restricted to only two groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes